CLINICAL TRIAL: NCT01644331
Title: The Targeting Acute Congestion With Tolvaptan In Congestive Heart Failure Study
Brief Title: Targeting Acute Congestion With Tolvaptan in Congestive Heart Failure
Acronym: TACTICS-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00037557
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure; Dyspnea
MeSH Terms: conditions — Heart Failure; Dyspnea | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tolvaptan (Experimental): Fixed-dose IV furosemide (1 x total daily oral dose given intravenously in divided doses Q12 hours OR 40 mg IV Q12 hours, whichever is greater) + oral Tolvaptan (given at 0, 24 and 48 hours)
  Interventions: Drug: Tolvaptan
- Placebo (Placebo Comparator): Fixed-dose IV furosemide (1 x total daily oral dose given intravenously in divided doses Q12 hours OR 40 mg IV Q12 hours, whichever is greater) + oral placebo (given at 0, 24 and 48 hours)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolvaptan — IV furosemide plusTolvaptan (given at 0, 24 and 48 hours)
  Other Names: Samsca
  Arms: Tolvaptan
Drug: Placebo — IV furosemide plus oral placebo (given at 0, 24 and 48 hours)
  Arms: Placebo

SUMMARY:
The primary objective of this study is to compare the effects of oral Tolvaptan vs. placebo as an adjunct to fixed dose IV furosemide on dyspnea relief in patients with acute decompensated heart failure

The primary hypothesis is that the addition of oral Tolvaptan to fixed dose furosemide will be more effective at relieving dyspnea than fixed dose furosemide alone

DETAILED DESCRIPTION:
This study will be a randomized, double blind, placebo controlled, multi-center clinical trial of patients with signs and symptoms consistent with AHF within 24 hours of presentation at Emergency Department. A total of approximately 250 patients will be enrolled in the trial.

Patients will be randomized in a 1:1 ratio to either of 2 treatment regimens:

* Fixed-dose IV furosemide (1 x total daily oral dose given intravenously in divided doses Q12 hours OR 40 mg IV Q12 hours, whichever is greater) + oral Tolvaptan (given at 0, 24 and 48 hours)
* Fixed-dose IV furosemide (1 x total daily oral dose given intravenously in divided doses Q12 hours OR 40 mg IV Q12 hours, whichever is greater) + oral placebo (given at 0, 24 and 48 hours)

The study treatment regimen will be administered from randomization through 48 hours, at which point Tolvaptan/placebo will be discontinued and all diuretic treatment will be adjusted at the treating physician's discretion.

The primary endpoint will be the proportion of patients with at least moderate improvement in dyspnea by Likert scale at both 8 AND 24 hours AND without the need for escalation of therapy due to worsening heart failure (rescue therapy) or death within 24 hours.

Patients will be followed daily for the duration of hospitalization or for 7 days (whichever is shortest).

All patients will have Day 30 follow up phone contact for assessment of vital status and interval hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Daily oral dose of furosemide between ≥ 40 mg(or equivalent)
* Identified within 24 hours of presentation, defined for purposes of this study as the time of initial dose of intravenous loop diuretic
* Prior clinical HF diagnosis that was treated with oral loop diuretics for at least 1 month
* Admission for acute decompensated Heart Failure (HF) as determined by

  * dyspnea at rest or with minimal exertion
  * Brain Natriuretic Peptide (BNP) > 400 or NTproBNP > 2000 pg/mL

AND at least one of the following additional signs and symptoms:

* Orthopnea
* Peripheral edema
* Elevated JVP (Jugular Venous Pressure)
* Pulmonary rales
* Congestion on Chest X-ray
* No plan for revascularization, cardiac transplant, of ventricular assist device implantation, or other cardiac surgery within 60 days of randomization
* Signed informed consent

Exclusion Criteria:

* Serum Na > 140 meq/L
* Received IV vasoactive treatment or ultra-filtration therapy for HF since initial presentation
* Treatment plan during current hospitalization includes IV vasoactive treatment or ultra-filtration for HF
* Systolic Blood Pressure (SBP)<90mmHg
* Serum-Cr>3.5mg/dl or currently undergoing renal replacement therapy

  . Known underlying liver disease
* Hemodynamically significant arrhythmias
* ACS(Acute coronary syndrome) within 4 weeks prior to study entry
* Active myocarditis
* Hypertrophic obstructive, restrictive, constrictive cardiomyopathy
* Severe stenotic valvular disease
* Complex congenital heart disease
* Constrictive pericarditis
* Clinical evidence of digoxin toxicity
* Need for mechanical hemodynamic support
* Terminal illness (other than heart failure) with expected survival time of less than 1 year
* History of adverse reaction to Tolvaptan
* Enrollment or planned enrollment in another randomized clinical trial during this hospitalization
* Pregnant or breast-feeding
* Inability to comply with planned study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2012-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Felker, MD, Principal Investigator — Duke Clinical Research Institute
Locations (18):
- United States (18):
  - University of Colorado at Denver and Health Sciences Center, Aurora, Colorado
  - Emory University School of Medicine, Atlanta, Georgia
  - Northeast Georgia Heart Center, Gainesville, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - University of Chicago, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Novant Health Heart and Vascular, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Grand View - Lehigh Valley Health Services, Sellersville, Pennsylvania
  - UT Southwestern Medical center, Dallas, Texas
  - Inova Heart and Vascular Institute, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided.

REFERENCES:
- [Derived] Felker GM, Mentz RJ, Cole RT, Adams KF, Egnaczyk GF, Fiuzat M, Patel CB, Echols M, Khouri MG, Tauras JM, Gupta D, Monds P, Roberts R, O'Connor CM. Efficacy and Safety of Tolvaptan in Patients Hospitalized With Acute Heart Failure. J Am Coll Cardiol. 2017 Mar 21;69(11):1399-1406. doi: 10.1016/j.jacc.2016.09.004. Epub 2016 Sep 18. PMID 27654854

RESULTS

PARTICIPANT FLOW:
Groups:
- Tolvaptan: IV furosemide (1 x oral dose given IV in Q12 hours divided doses or 40 mg IV Q12 hours, whichever is greater) plus oral Tolvaptan (given at 0, 12, 24 and 48 hours)
  Tolvaptan: Tolvaptan (given at 0, 12, 24 and 48 hours)
- Placebo: IV furosemide (1 x oral dose given IV Q12 divided doses or 40mg IV Q12 hours, whichever is greater) plus oral placebo (given at O, 24, 48 hours)
  Placebo: IV furosemide (1 x oral dose given IV in Q12 hours divided doses) plus oral placebo (given at 0, 12, 24 and 48 hours)
Period: Overall Study
Arm/Group | Tolvaptan | Placebo
Started | 129 | 128
Completed | 118 | 118
Not Completed | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolvaptan | Placebo | Total
Number analyzed (Participants) | 129 | 128 | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.42 (12.9) | 62.97 (15.7) | 64.70 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 42 | 86
  Male | 85 | 86 | 171
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 129 | 128 | 257

OUTCOME MEASURES:

1. Primary Outcome: Dyspnea Improvement Measured by Likert Scale at 8 and 24 Hours
Description: The number of patients with at least moderate improvement (as reported by patient) in dyspnea Likert scale at both 8 AND 24 hours AND without the need for escalation of therapy due to worsening heart failure (rescue therapy) or death within 24 hours.
Time Frame: 8 and 24 hours
Population: Baseline population
Measure: Count of Participants; unit: Participants
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 129 | 128
Participants | 20 | 26
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; Test type: Superiority or Other; p = 0.315, Chi-squared

2. Secondary Outcome: Renal Function
Description: Change in Serum creatinine from baseline to 24, 48 and 72 hours
Time Frame: 0, 24, 48 and 72 hours
Population: Baseline population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 129 | 128
mg/dL
  24 hours | 0.13 (0.4) | 0.04 (0.3)
  48 hours | 0.10 (0.4) | 0.05 (0.4)
  72 hours | 0.03 (0.6) | 0.06 (0.4)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; This is a repeated measures analysis so all rows (visits) are taken into account; Test type: Superiority or Other; p = 0.021, Mixed Models Analysis; Slope = 0.19, 95% CI 2-sided [0.03 to 0.34]

3. Secondary Outcome: Weight Loss
Description: Change in body weight from baseline to 24, 48, and 72 hours
Time Frame: 0, 24, 48, and 72 hours
Population: Baseline population
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 129 | 128
lbs
  24 hours | -4.41 (6.6) | -1.16 (13.2)
  48 hours | -6.11 (7.4) | -3.46 (6.3)
  72 hours | -8.19 (9.7) | -5.53 (7.0)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; This a repeated measure analysis so all rows (visits) are taken into account; Test type: Superiority or Other; p = 0.430, Mixed Models Analysis; Slope = 0.99, 95% CI 2-sided [-1.47 to 3.44]

4. Secondary Outcome: Fluid Loss
Description: Change from baseline fluid balance at 24, 48, and 72 hours
Time Frame: 0, 24, 48, and 72 hours
Population: baseline population
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 129 | 128
mL
  24 hours | -2182.25 (1844.4) | -1541.48 (1524.5)
  48 hours | -1948.01 (1635.6) | -1419.09 (1378.6)
  72 hours | -1757.09 (1670.4) | -1401.24 (1386.5)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; This is a repeated measures analysis so all rows (visits) are taken into account; Test type: Superiority or Other; p = 0.157, Mixed Models Analysis; Slope = -493.21, 95% CI 2-sided [-1176.96 to 190.55]

5. Secondary Outcome: Dyspnea Likert
Description: Number of patients that experience moderate or greater improvement (patient reported) in dyspnea by 7 point Likert scale at 48 and 72 hours
Time Frame: 48 and 72 hours
Population: baseline population
Measure: Count of Participants; unit: Participants
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 129 | 128
Participants
  48 hours | 88 | 74
  72 hours | 69 | 48
Statistical Analysis 1: Comparison: Placebo; This is a repeated measures analysis so all rows (visits) are taken into account; Test type: Superiority or Other; p = 0.206, Chi-squared

6. Secondary Outcome: Hospital Stay
Description: Total days spent in hospital from baseline until discharge or death
Time Frame: 7 days
Population: baseline population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 129 | 128
days | 6.46 (5.9) | 7.35 (7.0)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; Test type: Superiority or Other; p = 0.334, Log Rank; Kaplan Meier = 0.98, 95% CI 2-sided [0.96 to 0.99]

7. Secondary Outcome: Worsening or Persistent Heart Failure or Death
Description: Number of patients with worsening heart failure or death
Time Frame: 72 hrs
Population: baseline population
Measure: Count of Participants; unit: Participants
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 129 | 128
Participants | 54 | 60
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; Test type: Superiority or Other; p = 0.148, Chi-squared

8. Secondary Outcome: Over-diuresis
Description: clinical evidence of volume depletion requiring intervention other than holding diuretics during the 72 hours after randomization
Time Frame: 72 hours
Population: baseline population
Measure: Count of Participants; unit: Participants
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 129 | 128
Participants | 7 | 3
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; Test type: Superiority or Other; p = 0.334, Chi-squared

9. Secondary Outcome: Serum Sodium
Description: Change in serum sodium from baseline to 24, 48, and 72 hours
Time Frame: 0, 24, 48, and 72 hours
Population: baseline population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 129 | 128
mmol/L
  24 hours | 3.18 (3.3) | 0.23 (2.5)
  48 hours | 3.34 (3.7) | -0.24 (2.8)
  72 hours | 2.84 (3.9) | -0.44 (2.9)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; This is a repeated measures analysis so all rows (visits) are taken into account; Test type: Superiority or Other; p = 0.241, Mixed Models Analysis; Slope = -0.67, 95% CI 2-sided [-1.79 to 0.45]

10. Secondary Outcome: Dyspnea 11 Point NRS
Description: Change in NRS for assessment of dyspnea from baseline to 24, 48, and 72 hours (scale ranges from 0-No difficulty breathing to 10-Difficulty as bad as you can imagine)
Time Frame: 0, 24, 48, and 72 hours
Population: baseline population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 129 | 128
units on a scale
  24 hours | -2.20 (2.5) | -1.84 (2.1)
  48 hours | -2.85 (2.7) | -2.29 (2.3)
  72 hours | -3.07 (3.0) | -2.42 (2.4)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; This is a repeated measures analysis so all rows (visits) are taken into account; Test type: Superiority or Other; p = 0.303, Mixed Models Analysis; Slope = 0.28, 95% CI 2-sided [-0.26 to 0.82]

11. Secondary Outcome: Freedom From Congestion
Description: Jugular Venous Pressure (JVP) < 8 cm, no orthopnea, trace peripheral edema or less, and will be assessed at 24, 48, and 72 hours
Time Frame: 24, 48, and 72 hours
Population: baseline population
Measure: Count of Participants; unit: Participants
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 129 | 128
Participants
  24 hours | 9 | 12
  48 hours | 24 | 20
  72 hours | 27 | 17
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; Test type: Superiority or Other; p = 0.471, Chi-squared — 24 hours
Statistical Analysis 2: Comparison: Tolvaptan vs Placebo; Test type: Superiority or Other; p = 0.585, Chi-squared — 48 hrs
Statistical Analysis 3: Comparison: Tolvaptan; Test type: Superiority or Other; p = 0.120, Chi-squared — 72 hrs

12. Secondary Outcome: Development of Worsening Renal Function
Description: increase in serum creatinine ≥ 0.3mg/dl from randomization at any time point during 72 hours after randomization
Time Frame: 72 hours
Population: baseline population
Measure: Count of Participants; unit: Participants
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 129 | 128
Participants | 50 | 34
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; Test type: Superiority or Other; p = 0.037, Chi-squared

13. Secondary Outcome: Days Hospitalized or Deceased
Description: Total days hospitalized or deceased during the 30 days after randomization
Time Frame: 30 days
Population: baseline population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 129 | 128
days | 10.19 (10.9) | 11.69 (11.7)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; Test type: Superiority or Other; p = 0.373, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: All Cause Death or Rehospitalization
Description: All cause death or rehospitalization (to include unscheduled clinic visits or ED visits) at 30 days (Kaplan-Meier and 95% confidence interval)
Time Frame: 30 days
Population: baseline population
Measure: Mean (95% Confidence Interval); unit: proportion of participants
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 129 | 128
proportion of participants | 0.33 [0.25 to 0.42] | 0.29 [0.22 to 0.38]
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; Test type: Superiority or Other; p = 0.709, Log Rank; Kaplan Meier = 0.26, 95% CI 2-sided [0.21 to 0.32]

ADVERSE EVENTS:
Time Frame: Serious adverse events occurring from randomization through day 7 or discharge (whichever occurred first)
Arm/Group | Tolvaptan | Placebo
Serious Adverse Events (participants affected / at risk) | 8/129 | 2/128
Other Adverse Events (participants affected / at risk) | 101/129 | 107/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolvaptan (N=129) | Placebo (N=128)
Blood Sodium Increase (Renal and urinary disorders) | 1 (1) | 0 (0)
Epistaxis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 0 (0)
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Hyponatraemia (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolvaptan (N=129) | Placebo (N=128)
Atrial Fibrillation (Cardiac disorders) | 13 (13) | 19 (19)
Ventricular Tachycardia (Cardiac disorders) | 5 (5) | 7 (7)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute Renal Failure (Renal and urinary disorders) | 24 (24) | 15 (15)
Worsening Heart Failure (Cardiac disorders) | 49 (86) | 59 (106)
Death (Cardiac disorders) | 8 (8) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days